CLINICAL TRIAL: NCT06653166
Title: Retrospektive Analyse Von Patientendaten bezüglich Die notfallmässige Atemwegssicherungen Durch Den Rettungsdienst Zug (Airway Management Analysis in the Rescue Environment of the Emergency Service Zug) - Retrospective Analysis of Patient Data Regarding the Emergency Airway Management by the Rescue Service Zug
Brief Title: Retrospective Data Analysis With the Aim to Determine the Success Rate of Endotracheal Intubation in the First Attempt in the Zug Rescue Service With Various Airway Devices Already in Everyday Use
Acronym: AWARE
Status: Active, not recruiting | Type: Observational
Sponsor: Rettungsdienst Zug (Other Government)
Responsible Party: Sponsor
Other Study IDs: AWARE; 2024-02051 (Other: Ethics Committee Northwestern and Central Switzerland EKNZ)
Record Dates: First submitted 2024-10-18; First posted 2024-10-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Insufficiency; Intubation; Airway Management; Prehospital Airway Management in Patients With Cardiac Arrest; Prehospital Emergency Medical Services; Videolaryngoscopy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- videolaryngocopy with bougie (S Guide)
  Interventions: Device: bougie (S Guide); Device: videolaryngoscopy
- conventional laryngoscopy with bougie (S Guide)
  Interventions: Device: bougie (S Guide)
- videolaryngoscopy with introducer
  Interventions: Device: videolaryngoscopy
- conventional laryngoscopy with introducer

INTERVENTIONS:
Device: bougie (S Guide) — bougie (S Guide)
  Groups: conventional laryngoscopy with bougie (S Guide); videolaryngocopy with bougie (S Guide)
Device: videolaryngoscopy — videolaryngoscopy hyperangulated or Macintosh
  Groups: videolaryngocopy with bougie (S Guide); videolaryngoscopy with introducer

SUMMARY:
Airway management is a critical procedure in emergency medicine, especially endotracheal intubation, which can be life-saving. Various techniques, such as video laryngoscopes and conventional laryngoscopes, are used, with success depending on first-pass success. The aim of this retrospective data analysis is to determine the success rate of endotracheal intubation in the first attempt in the Zug Rescue Service between 01/20 and 01/25 with various airway management devices already used in everyday life. The individual complications should secondary with regard to frequency and category as well as possible risk factors. risk factors. The aim is to examine the data on airway management of patients who had to be intubated due to a critical illness (e.g. impaired oxygenation or ventilation, reduced vigilance, cardiovascular arrest, etc.). The data is continuously collected and evaluated by the RDZ as part of quality assurance.

DETAILED DESCRIPTION:
Securing the airway is a critical aspect of pre-hospital emergency medicine and a complex, often life-saving measure. Endotracheal intubation in particular is a key intervention to ensure adequate oxygenation and ventilation in critically ill or injured patients and to secure the airway. Despite the development of alternative airway devices, the endotracheal tube remains the gold standard in prehospital emergency care due to its reliability and ability to safely protect the airway from aspiration. The ability to perform rapid and successful endotracheal intubation is critical for healthcare professionals, as failure to secure the airway significantly increases mortality and morbidity. Failure to intubate the trachea on the first attempt (lack of first-pass success) occurs in up to 20% of tracheal intubations in the emergency department or intensive care unit and up to 40% of prehospital intubations and is associated with an increased risk of severe hypoxemia, aspiration, cardiac arrest and death. Given the often challenging conditions in the prehospital environment - such as limited space, suboptimal lighting and time pressure - mastering this technique becomes even more important. The airway should therefore be secured under the best possible conditions and with the aid of appropriate airway adjuncts. Despite advances, the optimal choice of laryngoscope and supportive devices remains a controversial topic in clinical practice with recommendations for the primary use of a video laryngoscope with a Macintosh-like blade in emergency medicine. Commonly used approaches to airway management include: the hyperangulated video laryngoscope, the video laryngoscope with Macintosh blade, the conventional laryngoscope, each in combination with a stylet or bougie. Each of these methods offers specific advantages and disadvantages that may be relevant in different clinical scenarios. In previous studies under everyday conditions and in simulations, video laryngoscopy showed mixed results compared to conventional laryngoscopy in terms of first-pass success (especially in experienced users) with a trend towards increased success rates for the first intubation attempt with video laryngoscopy and a better view of the glottis. The hyperangulated video laryngoscope promises an improved view of the glottis, especially in difficult airways, while the video laryngoscope with Macintosh blade bridges the gap between conventional and video-assisted laryngoscopy. The conventional laryngoscope is still widely used. The respective laryngoscopes are often supplemented by the use of a guide rod or a bougie (tube introducer) to facilitate intubation. Some of the comparative studies conducted to date have shown a trend towards better first-pass success using a bougie, but were also inconclusive. Despite numerous studies on individual aspects of these aids, a comparison of the methods in combination in real prehospital situations is still lacking. In addition, the data regarding first-pass success in endotracheal intubation is unclear when comparing medical and non-medical personnel - some studies showed no differences, while others showed a higher success rate for emergency medical personnel. Our retrospective study aims to close these gaps in knowledge by systematically examining the success rates, number of attempts to successful intubation, complication rates and ease of use of each method. The purpose of this data analysis is to develop evidence-based recommendations for the choice of the optimal airway adjunct and thus improve patient safety and the efficiency of prehospital airway management standards, thereby reducing mortality. The prehospital and clinical data already collected as part of the internal quality management of the emergency medical services offers the opportunity to determine the incidence of the important first-pass success with various airway devices and to record previously reported complications and incidents by evaluating the internal quality management system that has already been in operation for many years.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who have had their airway secured by endotracheal intubation by RDZ staff

Exclusion Criteria:

* Existence of a documented refusal.
* Age < 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim is to examine the data on airway management in the Zug Rescue Service who had to be intubated due to a critical illness (e.g. oxygenation or ventilation disorder, reduced vigilance, cardiovascular arrest, etc.). The data is continuously collected and evaluated by the RDZ as part of quality assurance.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Success rate (first pass success) with Video laryngoscope with Macintosh blade "C-MAC" used in the Zug rescue service | January 2020 to January 2025
Success rate (first pass success) with the hyperangulated video laryngoscope "D-BLADE" in the Zug rescue service | January 2020 to January 2025
Success rate (first pass success) with Conventional laryngoscope in the Zug rescue service | January 2020 to January 2025
Success rate (first pass success) with Surgical airway protection in the Zug rescue service | January 2020 to January 2025
Success rate (first pass success) with the Bougie/tube introducer in the Zug rescue service | January 2020 to January 2025
Success rate (first pass success) with the Stylet/guide rod in the Zug rescue service | January 2020 to January 2025

SECONDARY OUTCOMES:
Incidence of mechanical damage | January 2020 to January 2025
Incidence of airways retrospectively assessed as definitively difficult | January 2020 to January 2025
  proportion of "definitive difficult airway" to "anticipated difficult airway" and "unanticipated difficult airway"
Portion of Medical/non-medical occupational patients | January 2020 to January 2025
Incidence of drop in saturation SpO2 <90% | January 2020 to January 2025
Correlation of succes rate and years of clinical experience of the intubator | January 2020 to January 2025
Proportion of day or night shift on intubations with first pass effect | January 2020 to January 2025
Patient demographics (median age, proportion of gender) | January 2020 to January 2025
Reason for initiating resuscitation/DAI | January 2020 to January 2025

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Florian Scherr, MD, Principal Investigator — Rettungsdienst Zug
Locations (1):
- Rettungsdienst Zug, Zug, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brinkmann F, Cajoeri G, Sahli SD, Buehler PK, Scherr BF. Airway management analysis in the rescue environment of the emergency service Zug: a retrospective real-world evaluation. Scand J Trauma Resusc Emerg Med. 2025 Oct 22;33(1):171. doi: 10.1186/s13049-025-01489-x. PMID 41126289